CLINICAL TRIAL: NCT06871878
Title: PeRsonAlised Community Based TelerehabIlitation Post StrokE to Increase Rehabilitation Time and Improve Motor Recovery: a Feasibility Study
Brief Title: Feasibility of a Physiotherapy Programme, with Integrated TelerehabIlitation to Increase Rehabilitation Time and Improve Motor Function
Acronym: PRACTISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: University of Glasgow (Other); University of Aberdeen (Other); University of Dundee (Other); The Stroke Association, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRACTISE; SA PG2S21\100006 (Other Grant/Funding Number: Stroke Association)
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Stroke Patients; Stroke
Keywords: Stroke; Physiotherapy; Exercise; TelerehabIlitation; Feasibility; Goal-Setting; Self-managment
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An assessor who will collect outcome measures will be blinded to the groups. This study has an intervention and a usual care arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment As Usual (No Intervention): Participants randomised to the control group will receive usual multi-disciplinary rehabilitation from their care team (e.g., physiotherapist, Occupational Therapists, Speech and Language Therapists) as per their NHS Health boards care plan.
- PRACTISE Physiotherapy (Experimental): The PRACTISE programme is a 16-week personalised physiotherapy programme, incorporating tele-rehabilitation, which aims to support individuals to achieve optimal dose of exercise to improve motor and functional outcomes after stroke. There are three core components to the intervention: goal setting, exercise and a supported self-management approach. PRACTISE comprises of nine therapist supported sessions: five in person, home-based rehabilitation sessions (weeks 1-4, two visits in week 1) and four telephone or video consultations (Near Me) (weeks 6, 8, 12 and 16), a simple self-management workbook (with space to record personal goals, action plans and progress) to develop skills for self-management, and a personalised online exercise programme delivered through the Giraffe platform five times per week.
  Interventions: Other: PRACTISE Physiotherapy Intervention

INTERVENTIONS:
Other: PRACTISE Physiotherapy Intervention — The PRACTISE programme is a 16-week personalised physiotherapy programme, incorporating tele-rehabilitation, which aims to support individuals to achieve optimal dose of exercise to improve motor and functional outcomes after stroke. There are three core components to the intervention: goal setting, exercise and a supported self-management approach. PRACTISE comprises of nine therapist supported sessions: five in person, home-based rehabilitation sessions (weeks 1-4, two visits in week 1) and four telephone or video consultations (Near Me) (weeks 6, 8, 12 and 16), a simple self-management workbook (with space to record personal goals, action plans and progress) to develop skills for self-management, and a personalised online exercise programme delivered through the Giraffe platform five times per week.
  Arms: PRACTISE Physiotherapy

SUMMARY:
About two thirds of people after stroke have some level of disability. Rehabilitation helps to reduce disability and supports people to return to a meaningful life. We know that the more rehabilitation you do especially, within the first six months after stroke, the better the outcome. However, rehabilitation services, especially in the community, are often lacking, non-specialist or provide only a limited number of therapy sessions. Recently national guidelines for care of people after stroke recommend that people receive up to three hours/day of therapy on at least five days/week. NHS services cannot provide this level of therapy so new ways to support people to increase the amount of therapy they do on their own is needed.

The aim of the research is to test a 16 week community, home-based physiotherapy programme to improve the amount of therapy exercise a stroke survivor does, therefore improving the outcome and reducing the level of disability.

Participants will be recruited as they transition from inpatient services to community physiotherapy. Participants will be randomised to either the control or intervention arm. Participants in the intervention arm will take part in a 16-week community, home-based physiotherapy programme. Within the 16-week intervention, participants will receive 5 home based and 4 remote appointments which will comprise of usual physiotherapy assessment and exercise prescription that incorporates 1) Personalised online exercise programme delivered through the Giraffe platform; 2) Goal setting and Action Planning (G-AP); and 3) Supported self-management approaches. Participants will receive an intervention workbook to support them with strategies to achieve their goals and build their self-management skills e.g. how to integrate therapy into their daily life, dealing with barriers, identifying social support networks.

Participants randomised to the control group will receive usual multi-disciplinary rehabilitation from their care team (e.g., physiotherapist, Occupational Therapists, Speech and Language Therapists) as per their NHS Health boards care plan.

The study will measure both feasibility outcomes associated with the implementing the study alongside clinical and wellbeing measures.

To test the feasibility of the study we will assess how many people agree to take part, complete the exercise sessions and complete the outcome measurements. We will also interview people affected by stroke, their significant others if appropriate, and therapists to get their views on the programme. We will do clinical assessments too at four time points across the study looking at walking ability, arm function, level of disability, confidence level, fatigue and quality of life.

DETAILED DESCRIPTION:
Stroke affects around 100,000 people in the UK each year, is the leading cause of disability and the fourth leading cause of death in the UK. The first six months after stroke is the optimum time for neuroplasticity and recovery and therefore a critical period for rehabilitation. Exercise post-stroke needs to be repetitive, task-specific and high-dose to optimise motor and functional recovery. The recent National Clinical Guideline for Stroke recommends patients should receive at least three hours a day of multidisciplinary therapy at least five days week. Delivering this dose of therapy in community settings is challenging (e.g., waiting lists, therapist availability) and around 40% of stroke survivors are discharged home without any further rehabilitation and thus receive sub-optimal levels of therapeutic rehabilitation. Subsequently, alternative models of rehabilitation are required and there is a

One approach is to empower stroke survivors to take control of their own personal rehabilitation needs outside of NHS appointments. Progressing individuals towards the volume of therapy recommended by National Clinical Guideline for Stroke for optimal recovery benefits. Therefore, the investigators are seeking to combine previous stroke based research, from distinct areas, notably, Tele-rehabilitation, goal setting and self-management.

The PRACTISE intervention is based upon the use of tele-rehabilitation (Giraffe platform) incorporating evidence-based behavioural change techniques, with the addition of an evidence-based approach to support patients to set and pursue their personal goals (the Goal setting and Action Planning framework) and support for therapists to build trusted and supportive relationships for self-management (IMPETUS study).

Tele-rehabilitation, recommended by the new Stroke Guidelines, has the potential to address the issues of sub-optimal levels of therapeutic care by offering access to specialist services, reducing transport requirements/costs (therapist and patient), whilst allowing for personalisation services, increased dose of therapy and enhanced monitoring. The Telerehabilitation platform, Giraffe allows therapists to provide personalised, video-based exercise programmes and with an inbuilt exercise diary. Previous research has shown the feasibility of the Giraffe platform to augment upper-limb physiotherapy at the in-patient stage of stroke rehabilitation (30mins of additional therapy, up to five times/week) and found the intervention to be feasible, safe and acceptable to patients, carers and Physiotherapists.

Goal setting is a central and recommended component of stroke rehabilitation practice. The Goal setting and Action Planning (G-AP) framework is a theory- and evidence-based method, developed by one of our team, to support stroke survivors to consider, plan, and work towards their goals collaboratively with rehabilitation staff. Evaluations of G-AP in community stroke rehabilitation settings found it was acceptable to staff and people in their care, feasible to implement in practice and helpful in the setting and pursuit of person-centred goals.

Supported self-management is advocated for within national clinical guidelines and current stroke policies. It's an approach designed to help stroke survivors to regain their confidence to manage the impact of their stroke and live their lives well after a stroke. The IMPETUS study showed that supported self-management helps to improve stroke survivor's quality of life, confidence, independence and helps people to adopt lifestyle changes that reduce their risk of secondary stroke. Within PRACTISE, supported self-management is a collaborative discussion and mutual understanding between physiotherapist and participant to help people to develop the skills and confidence to self-manage well. Conversations with therapists will be supplemented with educational awareness components via a participant workbook that will support the participant with strategies to achieve their goals and build their self-management skills e.g. how to integrate therapy into their daily life, dealing with barriers, identifying social support networks.

The ultimate aim of this research is to determine if a personalised, goal-based, physiotherapy programme, with integrated tele-rehabilitation, to improve motor and functional outcomes in the first six months after stroke (PRACTISE), is clinically and cost effective compared to usual care. Prior to undertaking a definitive randomised controlled trial (RCT) this feasibility study will explore uncertainties about the intervention and trial.

ELIGIBILITY:
1. Individuals who have experienced a stroke.

   Inclusion criteria:
   * Over 16 years old
   * Within two months of first stroke
   * Requiring community physiotherapy and discharged home from in-patient care
   * Scores 2-4 on the modified Rankin Score on discharge
   * Able to use a computer/tablet or mobile phone with/without help from carers' (participants who lack digital connectivity skills/ Products will be assisted through AbilityNet)
   * Able to understand/communicate in English
   * Capacity to provide informed consent

   Exclusion criteria:
   * Participating in another physical interventional research study
   * Discharged to a nursing home or other long-term care facility
   * Absolute contra-indication to exercise
2. Carers or family members of individuals who have experienced a stroke.

   Inclusion criteria:
   * Significant other/carer of an individual who is part of the PRACTISE study either as a control participant or as an intervention participant
   * Over the age of 16 years
   * Able to join and contribute to an interview, either in-person or via a video conference platform, in English.
3. Treating physiotherapist who will deliver the PRACTISE intervention.

Inclusion criteria:

* UK-based Physiotherapist who has delivered the PRACTISE intervention
* Able to join and contribute to an interview via video conference platform or in person
* Over the age of 18 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Base line, week 8, week 16 and week 24 (follow up)
  The main aim of the Canadian Occupational Performance Measure is to identify occupational performance problems, concerns and issues of participants (wants to do, needs to do or is expected to do, but can't do, doesn't do or isn't satisfied with the way they do it). Through a discussion, participant identifies up to five problems they face in self-care, productivity and leisure. They then prioritise the activities and rate their current level of performance and satisfaction with each. The COPM is generally a reliable, valid, and acceptable tool for researchers with satisfactory test-retest reliability specifically in stroke. COPM results will be given to physiotherapist of intervention participant. This will allow discussion between the participant and physiotherapist to agree specific, and meaningful goals using the G-AP framework.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | Base line, week 8, week 16 and week 24 (follow up)
  The Action Research Arm Test is a 19-item physical measure to assess upper extremity performance (coordination, dexterity and functioning) in stroke recovery. It comprises 4 sub-tests (grasp, grip, pinch, and gross arm movement). Within each sub-test, assessments are arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Item scored on a four-point scale from 0 (can do no part of the test) to 3 (performs the test normally).
Motricity Index | Base line, week 8, week 16 and week 24 (follow up)
  Motricity Index assesses motor impairment and muscle strength of the upper and lower limbs and involves three upper limb activities; shoulder abduction, elbow flexion and pinch grip and three lower limbs; hip extension, knee extension and ankle dorsiflexion.
Timed Up and Go test | Base line, week 8, week 16 and week 24 (follow up)
  Timed up and go test assesses mobility, balance, walking ability, and fall risk. The participant stands from a chair, walks 3 metres at a comfortable pace, turns around, walks back to the chair and sits down. The time to complete the test is recorded and walking aids are used as required. The test will be conducted three times with the average score being calculated and used as the final measure.
The Barthel Index | Base line, week 8, week 16 and week 24 (follow up)
  The Barthel Index is a patient reported outcome and measures the extent to which somebody can function independently and has mobility in their activities of daily living. Activities of daily living measured include feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Each activity is scored out of 10, with a maximum of score 100.
The Stroke Specific Quality of Life questionnaire | Base line, week 8, week 16 and week 24 (follow up)
  The Stroke Specific Quality of Life questionnaire consists of 49 items each assessed on a 5-point scale. The domains covered include mobility, energy, work and productivity, mood, self-care, language, thinking and personality. Scores range from 49 to 245 with higher scores associated with higher quality of life.
EQ-5D-5L | Base line, week 8, week 16 and week 24 (follow up)
  EQ-5D-5L evaluates health-related quality of life with one question for each of the five dimensions mobility, self- care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The Eq-5D-5L also comprises a visual analogues scale that records the participants self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Fatigue Severity Scale | Base line, week 8, week 16 and week 24 (follow up)
  Fatigue Severity Scale is 9-item scale, that is self reported by participants. The scale measures the severity of fatigue and its effect on a person's life against 9 statements. Each item is scored on a scale of 1 (strongly disagree) -7 (strongly agree). Scores range from 9 to 63 with higher scores indicating more severe fatigue.
Stroke Self Efficacy Questionnaire | Base line, week 8, week 16 and week 24 (follow up)
  Stroke Self Efficacy Questionnaire is a self-report scale of self-efficacy post stroke that demonstrates good internal consistency and criterion validity. It is a 13-item patient reported outcome where participants rate their confidence with stated tasks from 0 not at all confident to 10 very confident. The SSEQ total score can potentially range from 0 to 130 with higher scores indicating higher levels of self-efficacy.
The Patient Experience of Treatment and Self-Management after Stroke | Baseline and week 16 only
  The Patient Experience of Treatment and Self-Management was developed to measure treatment burden in people with multi-morbidity and/or complex self-management regimens. However, it omits stroke-specific burdens. Therefore, the Patient Experience of Treatment and Self-Management after Stroke (PETS-STROKE) PETS-STROKE is a 34-item patient reported measure that captures the workload of healthcare and impact on wellbeing experienced by the stroke survivor.
Number of falls | Base line, week 8, week 16 and week 24 (follow up)
  The number of falls since the previous assessment will be self-reported, with a fall defined as 'an unexpected event in which the participant comes to rest on the ground, floor or lower'. As the intended outcome of the intervention is to increase functional activity this may increase risk of falls.
Caregiver strain index | Base line, week 8, week 16 and week 24 (follow up)
  Caregiver strain index This is a self report written questionnaire across 13-items which assesses the level of stress experienced by informal caregivers, answered with - Yes (2), Sometimes (1) or No (0). The maximum score is 26.

OTHER OUTCOMES:
Adherence/dose-response measure | Each therapy appointment
  Care delivered by physiotherapists, occupational therapists and speech and language therapists, for both CONTROL and INTERVENTION groups will be recorded by the therapist using a short checklist. This will include, date of appointment, duration of appointment, who the appointment was with (e.g., physiotherapist, speech and Language), and content via a checklist of usual care interventions. This will be completed for each therapy appointment
  Exercise diaries will be completed by participants either in the Giraffe platform (intervention) or paper (control). This information will be used to determine the weekly dose of exercise from which dose/response will be calculated for the clinical outcomes.
Feasibility outcomes measures | Recruitment, screening, baseline, week 8, week 16, week 24 (follow up)
  Data from screening, recruitment and follow-up logs will be used to generate realistic estimates of eligibility, recruitment, consent and follow-up rates, reasons for drop-out and adverse events. Outcome measure completion and missing data will also be recorded.
Intervention fidelity | Week 1, week 4, week 6, week 16
  To understand fidelity of PRACTISE, 20 audio recordings of PRACTISE sessions between a physiotherapist and a participant will be made. This will include 5 on session-1 (week 1), 5 on session-5 (week 4), 5 on session-6 (week 6) and 5 on session-9 (week 16). Physiotherapists will record these sessions via a Dictaphone. Equal representation will be sought across site locations.
Process evaluation | immediately after the intervention
  Interviews will be conducted to assess fidelity, acceptability and adherence of the study. Interviews will be conducted with:
  1. individuals who have had experienced a stroke,
  2. carer or significant others and
  3. treating physiotherapist.
  Interviews will be conducted after the 16-week intervention period for individuals who have experienced a stroke and for carers or significant others. Therapist interviews will be conducted when their involvement in the study is complete.
Economic outcome measures | From Baseline to week 16
  The economic analysis will focus on the feasibility and acceptability of collecting healthcare resource use and Quality of Life data required to conduct a full economic evaluation in a future trial. Item completion rates will be presented to assess data completeness. Data on the delivery of the PRACTISE intervention and usual care will be recorded by health care professionals during appointments with individuals who have experienced a stroke (described in dose response measure). Participants will be asked to record the aspects of their care in a record book on a weekly or as required basis during the 16-week period. This will include unplanned or urgent healthcare contacts in the last week, indicating who they saw, how, how many times, and if it was related to their stroke. The purchasing of any medication directly related to the stroke, purchase of exercise equipment to complete rehabilitation and digital devices used for tele-rehabiliton.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Paul, PhD, Principal Investigator — Glasgow Caledonian University

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publications will be available at request to other researchers.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be stored on One Drive for 10 years, after which it will be deleted and CRFs will be shredded as confidential waste.
Access Criteria: All IPD that underlie results in a publication will be available at request and stored on a Glasgow Caledonian University OneDrive account.

REFERENCES:
- [Background] Lyle RC. A performance test for assessment of upper limb function in physical rehabilitation treatment and research. Int J Rehabil Res. 1981;4(4):483-92. doi: 10.1097/00004356-198112000-00001. No abstract available. PMID 7333761
- [Background] Yang SY, Lin CY, Lee YC, Chang JH. The Canadian occupational performance measure for patients with stroke: a systematic review. J Phys Ther Sci. 2017 Mar;29(3):548-555. doi: 10.1589/jpts.29.548. Epub 2017 Mar 22. PMID 28356652
- [Background] Law M, Baptiste S, McColl M, Opzoomer A, Polatajko H, Pollock N. The Canadian occupational performance measure: an outcome measure for occupational therapy. Can J Occup Ther. 1990 Apr;57(2):82-7. doi: 10.1177/000841749005700207. PMID 10104738
- [Background] Brown SE, Scobbie L, Worrall L, Mc Menamin R, Brady MC. Access G-AP: development of an accessible goal setting and action planning resource for stroke survivors with aphasia. Disabil Rehabil. 2023 Jun;45(13):2107-2117. doi: 10.1080/09638288.2022.2085331. Epub 2022 Jun 11. PMID 35695078
- [Background] Bachmair EM, Martin K, Aucott L, Dhaun N, Dures E, Emsley R, Gray SR, Kidd E, Kumar V, Lovell K, MacLennan G, McNamee P, Norrie J, Paul L, Packham J, Ralston SH, Siebert S, Wearden A, Macfarlane G, Basu N; LIFT study group. Remotely delivered cognitive behavioural and personalised exercise interventions for fatigue severity and impact in inflammatory rheumatic diseases (LIFT): a multicentre, randomised, controlled, open-label, parallel-group trial. Lancet Rheumatol. 2022 Jun 27;4(8):e534-e545. doi: 10.1016/S2665-9913(22)00156-4. eCollection 2022 Aug. PMID 36388001
- [Background] Scobbie L, Duncan EAS, Brady MC, Thomson K, Wyke S. Facilitators and "deal breakers": a mixed methods study investigating implementation of the Goal setting and action planning (G-AP) framework in community rehabilitation teams. BMC Health Serv Res. 2020 Aug 25;20(1):791. doi: 10.1186/s12913-020-05651-2. PMID 32843039
- [Background] Scobbie L, McLean D, Dixon D, Duncan E, Wyke S. Implementing a framework for goal setting in community based stroke rehabilitation: a process evaluation. BMC Health Serv Res. 2013 May 24;13:190. doi: 10.1186/1472-6963-13-190. PMID 23705824
- [Background] Scobbie L, Dixon D, Wyke S. Goal setting and action planning in the rehabilitation setting: development of a theoretically informed practice framework. Clin Rehabil. 2011 May;25(5):468-82. doi: 10.1177/0269215510389198. Epub 2010 Dec 3. PMID 21131335
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Alhusayni AI, Cowey ES, Coulter E, Barber M, Paul L. Personalised Online Upper-Limb Physiotherapy for Stroke Survivors during the Inpatient Phase: A Feasibility Study. Healthcare (Basel). 2023 Sep 19;11(18):2582. doi: 10.3390/healthcare11182582. PMID 37761779
- [Background] Paul L, Renfrew L, Freeman J, Murray H, Weller B, Mattison P, McConnachie A, Heggie R, Wu O, Coulter EH. Web-based physiotherapy for people affected by multiple sclerosis: a single blind, randomized controlled feasibility study. Clin Rehabil. 2019 Mar;33(3):473-484. doi: 10.1177/0269215518817080. Epub 2018 Dec 4. PMID 30514108
- [Background] Rintala A, Paivarinne V, Hakala S, Paltamaa J, Heinonen A, Karvanen J, Sjogren T. Effectiveness of Technology-Based Distance Physical Rehabilitation Interventions for Improving Physical Functioning in Stroke: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2019 Jul;100(7):1339-1358. doi: 10.1016/j.apmr.2018.11.007. Epub 2018 Dec 6. PMID 30529323
- [Background] Appleby E, Gill ST, Hayes LK, Walker TL, Walsh M, Kumar S. Effectiveness of telerehabilitation in the management of adults with stroke: A systematic review. PLoS One. 2019 Nov 12;14(11):e0225150. doi: 10.1371/journal.pone.0225150. eCollection 2019. PMID 31714924
- [Background] Wu D, Zhang H, Leng Y, Li K, Li S, Lo WLA. A bibliometric analysis of telerehabilitation services for patients with stroke. Front Neurol. 2023 Jan 9;13:1026867. doi: 10.3389/fneur.2022.1026867. eCollection 2022. PMID 36698904
- [Background] Laver KE, Adey-Wakeling Z, Crotty M, Lannin NA, George S, Sherrington C. Telerehabilitation services for stroke. Cochrane Database Syst Rev. 2020 Jan 31;1(1):CD010255. doi: 10.1002/14651858.CD010255.pub3. PMID 32002991
- [Background] Russell TG. Physical rehabilitation using telemedicine. J Telemed Telecare. 2007;13(5):217-20. doi: 10.1258/135763307781458886. PMID 17697506
- [Background] Klassen TD, Dukelow SP, Bayley MT, Benavente O, Hill MD, Krassioukov A, Liu-Ambrose T, Pooyania S, Poulin MJ, Schneeberg A, Yao J, Eng JJ. Higher Doses Improve Walking Recovery During Stroke Inpatient Rehabilitation. Stroke. 2020 Sep;51(9):2639-2648. doi: 10.1161/STROKEAHA.120.029245. Epub 2020 Aug 19. PMID 32811378
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Background] Lee KB, Lim SH, Kim KH, Kim KJ, Kim YR, Chang WN, Yeom JW, Kim YD, Hwang BY. Six-month functional recovery of stroke patients: a multi-time-point study. Int J Rehabil Res. 2015 Jun;38(2):173-80. doi: 10.1097/MRR.0000000000000108. PMID 25603539
- See also: Stroke rehabilitation in adults NICE guideline Published: 18 October 2023 — https://www.nice.org.uk/guidance/ng236/resources/stroke-rehabilitation-in-adults-pdf-66143899492549